CLINICAL TRIAL: NCT01769118
Title: The Influences of Caffeine on HRV of Preterm Infants
Brief Title: The Influences of Caffeine on Heart Rate Variability of Preterm Infants
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, wamir, Dr., Rambam Health Care Campus
Other Study IDs: 0442-12
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Autonomic Nervous System
Keywords: Autonomic nervous system
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Caffeine: caffeine will be given according to clinical judgment
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Caffeine will be given according to departmental protocol

SUMMARY:
Caffeine has a stimulatory effect on the ANS. This has not yet been investigated in preterm infant who get caffeine before stopping ventilation. The investigators hypothesis is that this stimulatory effect may be characterized by HRV analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* infants born before 34 weeks gestation

Exclusion Criteria:

* sepsis
* congenital malformations

Ages: 25 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 25 preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 1 hour
  Heart rate, SD, SDNN, HF, LF, VLF, TP

CONTACTS AND LOCATIONS:
Locations (1):
- RMC, Haifa, Israel